CLINICAL TRIAL: NCT06333431
Title: The Effects of Glass Waterfall and White Noise on Pain, Anxiety and Physiological Parameters During Gastroscopy
Brief Title: Effects of WN and WF During Gastroscopy
Acronym: WF/WN_GCPY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Hasan Genç, Asistant Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WN/WF
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Misadventure During Endoscopic Examination
Keywords: white noise; glass waterfall; anxiety, pain; gastroscopy
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment experimental model using randomized pretest and posttest with control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glass Waterfall (Experimental): Except for the preparation the gastroscopy procedure takes approximately 20 minutes, patients will be asked to focus on portative glass waterfall during the procedure.
  Interventions: Device: Glass Waterfall group
- White Noise (Experimental): Except for the preparation of the patient for the procedure, since the gastroscopy procedure takes approximately 20 minutes, 20-minute white noise be listened using phone
  Interventions: Device: white noise group
- control group (No Intervention): Patients of the control group, will not receive any intervention except for applied routine hospital gastroscopy procedures.

INTERVENTIONS:
Device: Glass Waterfall group — Except for the preparation the gastroscopy procedure takes approximately 20 minutes, patients will be asked to focus on portative glass waterfall during the procedure.
  Arms: Glass Waterfall
Device: white noise group — Except for the preparation of the patient for the procedure, since the gastroscopy procedure takes approximately 20 minutes, 20-minute white noise be listened using phone
  Arms: White Noise

SUMMARY:
Background: Gastroscopy is an endoscopic procedure that allows examination of the upper gastrointestinal system, including the esophagus, stomach and duodenum. The procedure is a difficult and stressful diagnosis and treatment method for the patient. Problems such as stress, fear and pain experienced during endoscopy cause anxiety.

Purpose: To examine effects of glass waterfall and white noise on pain, anxiety and physiological parameters during gastroscopy Method: The population of the study consists of all patients who applied to Mardin Education and Research Hospital, Department of General Surgery, Endoscopy Unit and were scheduled for gastroscopy. The sample will be represented by 156 patients whose gastroscopy procedure is planned between the specified dates and who meet the criteria for inclusion in the sample. In calculating the sample of the study, power analysis was performed and it was found the effect size of 1.16, 95% power and 0.05% margin of error for this study, that a total of 156 individuals for the three groups and at 52 individuals for each group. Before gastroscopy procedure, the patients included in the study will be randomly divided into three groups: 52 glass waterfall group, 52 white noise group and 52 control group.

DETAILED DESCRIPTION:
Background: Gastroscopy is an endoscopic procedure that allows examination of the upper gastrointestinal system, including the esophagus, stomach and duodenum. The procedure is a difficult and stressful diagnosis and treatment method for the patient. Problems such as stress, fear and pain experienced during endoscopy cause anxiety.

Purpose: To examine effects of glass waterfall and white noise on pain, anxiety and physiological parameters during gastroscopy Method: The population of the study consists of all patients who will apply to Mardin Education and Research Hospital, Department of General Surgery, Endoscopy Unit and will be scheduled for gastroscopy. The sample will be represented by 156 patients whose gastroscopy procedure is planned between the specified dates and who meet the criteria for inclusion in the sample. In calculating the sample of the study, power analysis will be performed and it is found the effect size of 1.16, 95% power and 0.05% margin of error for this study, that a total of 156 individuals for the three groups and at 52 individuals for each group. Before gastroscopy procedure, the patients included in the study will be randomly divided into three groups: 52 glass waterfall group, 52 white noise group and 52 control group.

Data will be collected in the endoscopy unit on weekdays when the procedure is performed. All participants in the study will first fill out a patient identification form containing patient demographic information.

ELIGIBILITY:
Inclusion Criteria:

* 18 aged and over
* Written and verbal consent to participate in the study,
* Being conscious (person, place and time orientation),
* Undergoing gastroscopy for the first time

Exclusion Criteria:

* Having vision, hearing and communication problems
* Having any psychiatric and cognitive/mental mental health problems, disease (dementia, etc.),
* Diagnosed with visual, auditory and / or balance disorders,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-04-03 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | the fundamental characteristics of the patients will be filled in 15 minutes before the gastroscopy procedure
  This form, which will be created by the researcher; Patients' age, gender, education level, marital status, employment status, income level, chronic disease status, previous surgery, complaints about coming to the hospital, whether they would prefer the current method if they need to have gastroscopy again, It consists of a total of 10 questions.
Visual Analogue Scale (VAS) | Change from Baseline Visual Analogue Scale in 50 minutes
  This scale developed by Price (1983) will be used in the research to determine the level of tolerance, comfort and satisfaction. It is a scale in which the distance between the two ends with a minimum value of 0 on one end and a maximum value of 10 on the other end is measured with a 10 cm ruler. In this context; The patient is explained that there are two endpoints and that he is free to mark any place between them that fits the severity of his pain.
  The distance between the beginning of "no comfort, tolerance and satisfaction" and this point marked by the patient is measured and recorded in centimeters. It has been shown that the VAS is a valid tool for the measurement of psychological and health variables such as pain and satisfaction, which is widely used in clinical studies
State and Trait Anxiety Scale (STAI) | Change from Baseline The State and Trait Anxiety Scale in 50 minutes
  It is a self-assessment questionnaire developed by Spielberger et al. and consists of short assessments. The STAI includes 40 four-point Likert-type items ranging from "None" to "Completely". The validity and reliability of the STAI in Turkey were established by Öner and Le Compte. The STAI includes two separate scales, the State Anxiety Score (SAS) and the Trait Anxiety Score (TAS). The SAS requires the person to describe how they feel at a certain moment and under certain conditions and to respond by taking into account their feelings about the situation they are in. Higher scores indicate increased anxiety level. In the Turkish validity and reliability study, Cronbach's alpha reliability coefficients were between 0.83 and 0.87 for the TAS and between 0.94 and 0.96 for the SAS.
The Patient Observation Form | Change from Baseline The Patient Observation Form in 50 minutes
  This form will be created by the researcher based on the literature review, the physiological parameters (pulse (min), respiratory rate (min), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and oxygen saturation values (%)) of the patients before and after the procedure will be recorded the form. Researcher will has a automatic blood pressure monitor and a probe device for recording the variables in the endoscopy unit. While the patients' physiological parameters will being taken, a fully automatic blood pressure monitor will be used to measure blood pressure and pulse. To measure the respiratory rate, the patient placed his hand on his chest and his chest movements will be counted and recorded for one minute. Oxygen saturation level will be measured from the index finger with a probe device. Data will be collected by recording all parameters measurement values on a single form. The form will similar to forms commonly used in nursing research.
Pulse rate before and after gatroscopy procedure | Change from Baseline Pulse rate in 50 minutes
  60 to 100 beats per minute is normal. It will be recorded 15 minutes before and after the gastroscopy procedure
Respiratory rate before and after gatroscopy procedure | Change from Baseline Respiratory rate in 50 minutes
  12 to 18 breaths per minute is normal. It will be recorded 15 minutes before and after the gastroscopy procedure
Systolic and diastolic blood pressure before and after gatroscopy procedure | Change from Baseline Systolic and diastolic blood pressure in 50 minutes
  90/60 mm Hg to 120/80 mm Hg is normal. It will be recorded 15 minutes before and after the gastroscopy procedure
Oxygen saturation values before and after gatroscopy procedure | Change from Baseline Oxygen saturation values in 50 minutes
  Normal oxygen saturation usually ranges from 95 to 100%. It will be recorded 15 minutes before and after the gastroscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hasan GENC, PhD, Principal Investigator — Dicle University

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

REFERENCES:
- [Result] Utli H, Dogru BV. The Effect of Reiki on Anxiety, Stress, and Comfort Levels Before Gastrointestinal Endoscopy: A Randomized Sham-Controlled Trial. J Perianesth Nurs. 2023 Apr;38(2):297-304. doi: 10.1016/j.jopan.2022.08.010. Epub 2022 Oct 20. PMID 36272846
- [Result] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Result] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Result] Umezawa S, Higurashi T, Uchiyama S, Sakai E, Ohkubo H, Endo H, Nonaka T, Nakajima A. Visual distraction alone for the improvement of colonoscopy-related pain and satisfaction. World J Gastroenterol. 2015 Apr 21;21(15):4707-14. doi: 10.3748/wjg.v21.i15.4707. PMID 25914482
- [Result] Veldhuijzen G, Klaassen NJM, Van Wezel RJA, Drenth JPH, Van Esch AA. Virtual reality distraction for patients to relieve pain and discomfort during colonoscopy. Endosc Int Open. 2020 Jul;8(7):E959-E966. doi: 10.1055/a-1178-9289. Epub 2020 Jun 30. PMID 32626819
- [Result] Ilkkaya NK, Ustun FE, Sener EB, Kaya C, Ustun YB, Koksal E, Kocamanoglu IS, Ozkan F. The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. J Perianesth Nurs. 2014 Oct;29(5):418-26. doi: 10.1016/j.jopan.2014.05.008. PMID 25261145
- [Result] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- [Derived] Genc H, Tanriverdi S. The Effects of a Portative Glass Waterfall and a White Noise App On Pain, Anxiety, and Physiological Parameters During Gastroscopy. Pain Manag Nurs. 2025 Oct 22:S1524-9042(25)00288-7. doi: 10.1016/j.pmn.2025.10.001. Online ahead of print. PMID 41130873